CLINICAL TRIAL: NCT03134872
Title: A Phase III, Randomized, Open-Label, Multi-center Study of SHR-1210(Anti-PD-1 Antibody) in Combination With Pemetrexed and Carboplatin as First Line Therapy in Subjects With Advanced/Metastatic Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study of SHR-1210 in Combination With Pemetrexed and Carboplatin in Subjects With Non-squamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-303-NSCLC
Record Dates: First submitted 2017-04-25; First posted 2017-05-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Respiratory Tract Disease; Neoplasms by Site; Neoplasm, Bronchial; Carcinoma, Bronchogenic
Keywords: PD-1; PD-L1; SHR-1210; Carboplatin; Pemetrexed
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Respiratory Tract Diseases; Neoplasms by Site; Bronchial Neoplasms; Carcinoma, Bronchogenic | interventions — camrelizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210+Chemotherapy (Experimental): Subjects receive SHR-1210 200mg and pemetrexed 500 mg/m^2 and carboplatin AUC 5, administered as IV infusion on Day 1 of each 21-day cycle for 4-6 cycles followed by optional SHR-1210 200mg and pemetrexed 500 mg/m^2 every three weeks (Q3W) maintenance for the remainder of the study or until documented PD.
  Interventions: Biological: SHR-1210; Drug: Carboplatin; Drug: Pemetrexed
- Chemotherapy (Active Comparator): Subjects receive pemetrexed 500 mg/m^2 and carboplatin Area Under the Curve (AUC) 5, administered as IV infusion on Day 1 of each 21-day cycle for 4-6 cycles followed by optional pemetrexed 500 mg/m^2 every three weeks (Q3W) maintenance for the remainder of the study or until documented PD. If PD occurs, Subjects may be able to receive SHR-1210 Q3W for the remainder of the study or until documented PD.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.
  Arms: SHR-1210+Chemotherapy
Drug: Carboplatin — Carboplatin
Drug: Pemetrexed — Pemetrexed

SUMMARY:
SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody. This is a randomized,Phase III, multicenter ,open-label study designed to evaluate the safety and efficacy of SHR-1210 with carboplatin and pemetrexed versus carboplatin-pemetrexed in subjects who are chemotherapy naive and have Stage IIIB/IV non-squamous NSCLC.

The primary hypothesis is that SHR-1210 combined with carboplatin and pemetrexed prolongs Progression Free Survival (PFS) in per RECIST 1.1 by blinded independent central review (ITT population and population was indicated by high PD-L1 expression) compared to carboplatin and pemetrexed treatment .

DETAILED DESCRIPTION:
In this study, subjects will be randomly assigned to receive either carboplatin and pemetrexed for 4-6 cycles followed by pemetrexed maintenance until progression or unacceptable toxicity, OR receive SHR-1210 combined with carboplatin and pemetrexed chemotherapy for 4-6 cycles followed by pemetrexed maintenance with SHR-1210 until progression or unacceptable toxicity (SHR-1210 for a maximum of 2 years).

Subjects assigned to the chemotherapy arm will have the opportunity to crossover to receive SHR-1210 monotherapy once they experience progression of disease (PD) defined by RECIST 1.1 and meet all the crossover criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are chemotherapy naive and have Stage IIIB-IV non-squamous NSCLC.
* 2. Subjects should not have a previously detected sensitizing EGFR mutation or ALK fusion oncogene.
* 3. Fresh cutting or ≤6 months preservation specimens must be provided.
* 4. No prior systemic treatment. Subjects who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment free interval of at least 12 months from randomization since the last chemotherapy cycle.
* 5. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria;
* 6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* 7. Have a life expectancy of at least 3 months.
* 8. All baseline laboratory requirements will be assessed and should be obtained within 14 days prior to the first administration of study treatment.
* 9. Female Subjects of childbearing potential must have a negative serum pregnancy test within 3 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 180 days after the last dose of study treatment.
* 10. Male Subjects with a female partner(s) of child-bearing potential must be willing to use very efficient barrier methods of contraception for the course of the study through 180 days after the last dose of study treatment.
* 11. Subjects has voluntarily agreed to participate by giving written informed consent/assent for the trial. The subject may also provide consent/assent for Future Biomedical Research.

Exclusion Criteria:

* 1. Target Disease Exceptions

  1. Subjects with predominantly squamous cell histology NSCLC, or SCLC.
  2. Subjects with epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) translocation.
  3. Subjects with no measurable disease by CT or MRI per RECIST 1.1 criteria.
  4. Subjects with carcinomatous meningitis, or symptoms of spinal cord compression.
  5. Subjects with active CNS metastases are excluded.
  6. Subjects who can receive surgical resection or radical radiotherapy.
  7. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* 2. Medical History and Concurrent Diseases

  1. Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger, or not requiring systemic treatment are permitted to enroll.
  2. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
  3. Prior therapy with systemic immunostimulatory agents within 1 months of the first dose of trial treatment.
  4. Subjects are currently participating and receiving study therapy or had participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 half-value period life of the agent, before the first dose of trial treatment.
  5. Subjects who expected to require any other form of antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC).
  6. Subjects received major surgery or radiation therapy of > 30 Gy not to chest within 4 weeks of the first dose of study treatment, or radiation therapy of > 30 Gy to chest within 24 weeks of the first dose of study treatment, or radiation therapy of < 30 Gy to chest within 2 weeks of the first dose of study treatment, and had not recovered from the toxicity and/or complications of the most recent prior chemotherapy to Grade 1 or less (except alopecia or fatigue).
  7. Subjects with a history of interstitial lung disease, or other disease may interfere with the detection or treatment of suspected drug-related lung toxicity.
  8. Other active malignancy requiring concurrent intervention.
  9. Subjects with previous malignancies (except non-melanoma skin cancers, and thefollowing in situ cancers: bladder, endometrial, cervical/dysplasia) are excluded unless a complete remission was achieved at least 5 years prior to study entry.
  10. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
  11. Subjects with active pulmonary tuberculosis.
  12. Subjects have severe infections within 4 weeks of the first dose of study treatment.
  13. Subjects had or plan to have allogeneic bone marrow transplantation or solid organ transplant.
  14. Subjects had administration of a live, attenuated vaccine within 30 days of the first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study.
  15. Subjects with contraindications to platinum therapy.
* 3. Physical and Laboratory Test Findings

  1. Known history of testing positive for human immunodeficiency virus (HIV) or
  2. known acquired immunodeficiency syndrome (AIDS).
  3. Known history of active Hepatitis B or C.
  4. Subjects with severe pleural effusion, pericardial effusion, or ascites need repeated drainage.
* 4. History of severe hypersensitivity reactions to other monoclonal antibodies, or intravenous infusion, or carboplatin, or pemetrexed.
* 5. Subjects have known psychiatric or substance abuse disorder (including alcohol\smoking), or be regular user (including "recreational use") of any illicit drugs that would interfere with cooperation with the requirements of the trial.
* 6. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival in the intent-to-treat (ITT) population | up to 24 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.
Progression-Free Survival in the PD-L1-selected population | up to 24 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 24 months
  Determined using RECIST v1.1 criteria
Duration of Response Rate(DoR) | up to 24 months
  Determined using RECIST v1.1 criteria
Time To Progression (TTP) | up to 24 months
  Determined using RECIST v1.1 criteria
Disease Control Rate (DCR) | up to 24 months
  Determined using RECIST v1.1 criteria
Overall Survival | up to 24 months
  Defined as the time from randomization to death from any cause.
Number of Subjects with treatment-related adverse events (AEs) | up to 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Tongji University, Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou C, Chen G, Huang Y, Zhou J, Lin L, Feng J, Wang Z, Shu Y, Shi J, Hu Y, Wang Q, Cheng Y, Wu F, Chen J, Lin X, Wang Y, Huang J, Cui J, Cao L, Liu Y, Zhang Y, Pan Y, Zhao J, Wang L, Chang J, Chen Q, Ren X, Zhang W, Fan Y, He Z, Fang J, Gu K, Dong X, Jin F, Gao H, An G, Ding C, Jiang X, Xiong J, Zhou X, Hu S, Lu P, Liu A, Guo S, Huang J, Zhu C, Zhao J, Gao B, Chen Y, Hu C, Zhang J, Zhang H, Zhao H, Wang Z, Ma X, Shi W. Camrelizumab plus carboplatin and pemetrexed as first-line therapy for advanced non-squamous non-small-cell lung cancer: 5-year outcomes of the CameL randomized phase 3 study. J Immunother Cancer. 2024 Nov 27;12(11):e009240. doi: 10.1136/jitc-2024-009240. PMID 39608979
- [Derived] Zhou C, Chen G, Huang Y, Zhou J, Lin L, Feng J, Wang Z, Shu Y, Shi J, Hu Y, Wang Q, Cheng Y, Wu F, Chen J, Lin X, Wang Y, Huang J, Cui J, Cao L, Liu Y, Zhang Y, Pan Y, Zhao J, Wang L, Chang J, Chen Q, Ren X, Zhang W, Fan Y, He Z, Fang J, Gu K, Dong X, Jin F, Gao H, An G, Ding C, Jiang X, Xiong J, Zhou X, Hu S, Lu P, Liu A, Guo S, Huang J, Zhu C, Zhao J, Gao B, Chen Y, Hu C, Zhang J, Zhang H, Zhao H, Tai Y, Ma X, Shi W; CameL Study Group. Camrelizumab Plus Carboplatin and Pemetrexed as First-Line Treatment for Advanced Nonsquamous NSCLC: Extended Follow-Up of CameL Phase 3 Trial. J Thorac Oncol. 2023 May;18(5):628-639. doi: 10.1016/j.jtho.2022.12.017. Epub 2023 Jan 13. PMID 36646210
- [Derived] Wu F, Jiang T, Chen G, Huang Y, Zhou J, Lin L, Feng J, Wang Z, Shu Y, Shi J, Hu Y, Wang Q, Cheng Y, Chen J, Lin X, Wang Y, Huang J, Cui J, Cao L, Liu Y, Zhang Y, Pan Y, Zhao J, Wang L, Chang J, Chen Q, Ren X, Zhang W, Fan Y, He Z, Fang J, Gu K, Dong X, Zhang T, Shi W, Zou J, Bai X, Ren S, Zhou C; CameL Study Group. Multiplexed imaging of tumor immune microenvironmental markers in locally advanced or metastatic non-small-cell lung cancer characterizes the features of response to PD-1 blockade plus chemotherapy. Cancer Commun (Lond). 2022 Dec;42(12):1331-1346. doi: 10.1002/cac2.12383. Epub 2022 Nov 4. PMID 36331328
- [Derived] Xie Q, Zheng H, Su N, Li Q. Camrelizumab in patients with advanced non-squamous non-small cell lung cancer: a cost-effective analysis in China. BMJ Open. 2022 Aug 5;12(8):e061592. doi: 10.1136/bmjopen-2022-061592. PMID 36194670
- [Derived] Chen T, Xie R, Zhao Q, Cai H, Yang L. Cost-Utility Analysis of Camrelizumab Plus Chemotherapy Versus Chemotherapy Alone as a First-Line Treatment for Advanced Nonsquamous Non-Small Cell Lung Cancer in China. Front Oncol. 2022 Jul 22;12:746526. doi: 10.3389/fonc.2022.746526. eCollection 2022. PMID 35936702
- [Derived] Zhou C, Chen G, Huang Y, Zhou J, Lin L, Feng J, Wang Z, Shu Y, Shi J, Hu Y, Wang Q, Cheng Y, Wu F, Chen J, Lin X, Wang Y, Huang J, Cui J, Cao L, Liu Y, Zhang Y, Pan Y, Zhao J, Wang L, Chang J, Chen Q, Ren X, Zhang W, Fan Y, He Z, Fang J, Gu K, Dong X, Zhang T, Shi W, Zou J; CameL Study Group. Camrelizumab plus carboplatin and pemetrexed versus chemotherapy alone in chemotherapy-naive patients with advanced non-squamous non-small-cell lung cancer (CameL): a randomised, open-label, multicentre, phase 3 trial. Lancet Respir Med. 2021 Mar;9(3):305-314. doi: 10.1016/S2213-2600(20)30365-9. Epub 2020 Dec 18. PMID 33347829